CLINICAL TRIAL: NCT07290543
Title: Designing for Sustainability: Co-Designing and Testing the Efficacy of a Web-Based Toolkit to Improve Cancer-Related Emotional Distress and Anxiety for Rural Older Cancer Survivors
Brief Title: Web-Based Toolkit to Improve Cancer-Related Emotional Distress and Anxiety in Rural Older Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: NU 24CC20; NCI-2024-09384 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00222660; NU 24CC20 (Other: Northwestern University); P30CA060553 (NIH); R01NR021666 (NIH)
Record Dates: First submitted 2025-09-24; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Early Intervention, Educational; Educational Status; Methods; Interviews as Topic; Patient Navigation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study staff abstracting the data will be blinded to the participant's condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (Advisory board) (Experimental): Advisory board members complete small group workshops, interviews and surveys on study.
  Interventions: Other: Interview; Other: Survey Administration
- Arm II (CONNECT platform) (Experimental): Patients and their caregivers receive access to the CONNECT platform, which includes educational materials on distress management, guides to telehealth and personalized recommendations for resources. Patients and their caregivers complete a guided tutorial of the platform with a research assistant at the start of the intervention period, receive biweekly phone calls with the research assistant, for 20 minutes starting on 14 days to 2 months to review the four cancer-related management functions and receive a text message reminders to encourage use, every 2 weeks for 4 months.
  Interventions: Other: Educational Intervention; Other: Internet-Based Intervention; Other: Interview; Behavioral: Patient Navigation; Other: Survey Administration; Behavioral: Telephone-Based Intervention; Other: Text Message-Based Navigation Intervention
- Arm III (Educational brochure) (Active Comparator): Patients are mailed an educational brochure about distress management on study.
  Interventions: Other: Educational Intervention; Other: Interview; Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention — Receive educational materials on distress management and guides to telehealth
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm II (CONNECT platform)
Other: Educational Intervention — Receive written educational brochure about distress management
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm III (Educational brochure)
Other: Internet-Based Intervention — Receive access to CONNECT platform
  Arms: Arm II (CONNECT platform)
Other: Interview — Complete interview
Other: Interview — Complete small group workshop
  Arms: Arm I (Advisory board)
Behavioral: Patient Navigation — Receive personalized recommendations for resources
  Other Names: Patient Navigator Program
  Arms: Arm II (CONNECT platform)
Other: Survey Administration — Ancillary study
Behavioral: Telephone-Based Intervention — Complete calls with research assistant
  Arms: Arm II (CONNECT platform)
Other: Text Message-Based Navigation Intervention — Receive text message reminders
  Other Names: Automated Text Message-Based Navigation; Text Message-Based Navigation
  Arms: Arm II (CONNECT platform)

SUMMARY:
This clinical trial tests how well a web based toolkit works to improve cancer related emotional distress and anxiety in rural older cancer survivors. Rural older adults with cancer-related distress are particularly vulnerable to poorer mental health and cancer-related outcomes including increased difficulties identifying symptoms of anxiety, a reduced likelihood of knowing when to access mental health services, and a higher likelihood of having poorly managed CRD, even after receiving a psychosocial referral. The web based tool kit called CONNECT addresses digital literacy and supports for cancer-related distress management through interactive activities for setting up telehealth visits, accessing educational materials about cancer-related distress, and providing individualized mental health resource recommendations. Using CONNECT may improve cancer related emotional distress and anxiety in rural older cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Co-design Objective (Aim 1): Finalize the CONNECT digital tool design through qualitative co-design evaluations with stakeholders to prepare the intervention for efficacy testing.

II. Efficacy Objective (Aim 2): Evaluate the efficacy of the CONNECT digital tool in reducing cancer-related distress among rural cancer survivors and caregivers, as measured by the validated 23-item Cancer and Treatment Distress Scale (CTXD), in a randomized controlled trial.

III. Implementation Objective (Aim 3): Assess the feasibility and potential for scale-up of the CONNECT intervention in rural communities and healthcare settings through qualitative interviews.

SECONDARY OBJECTIVES:

I. Assess self-reported healthcare resource utilization over the 12-month study period. (Aim 2, Efficacy Testing)

II. Assess self-reported shared device use for accessing health-related information and services. (Aim 2, Efficacy Testing)

III. Assess self-reported telehealth utilization, including portal use, completed visits, and visit modality. (Aim 2, Efficacy Testing)

IV. Evaluate cancer survivors' unmet needs using a validated 35-item unmet needs survey. (Aim 2, Efficacy Testing)

V. Evaluate caregiver strain using the validated 13-item Caregiver Strain Index. (Aim 2, Efficacy Testing)

OUTLINE: Advisory board members are assigned to arm I, patients and their caregivers are randomized to arm II or III.

ARM I: Co-design / Advisory Board Arm (Non-randomized) Advisory board members participate in qualitative co-design activities to refine the CONNECT digital tool prior to efficacy testing. Activities include small-group workshops, interviews, field-testing, and surveys focused on usability, content relevance, and acceptability of the platform.

ARM II: Intervention (CONNECT) Arm: Participants receive access to the CONNECT digital platform, which includes educational materials on cancer-related distress management, guidance on telehealth use, and personalized recommendations for supportive resources. They complete a guided onboarding tutorial with a Study Team Member, receive up to four structured review sessions (20 minutes each) by phone or video, and get automated text message reminders every two weeks for four months to encourage engagement.

Control Arm: Participants receive usual care plus a mailed educational brochure about managing cancer-related distress. They do not receive access to the CONNECT platform or coaching sessions.

ARM III: Patients are mailed an educational brochure about distress management on study. AIM 3: Scale-up / Implementation Assessment A subsample of participants from Arms II and III will participate in exit interviews to assess potential implementation outcomes, sustainability, and barriers/facilitators for scaling CONNECT in rural communities and healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1: Invited by a member of the study team
* AIM 1: In the following or related field:

  * Healthcare professionals (physicians, nurses, pharmacists, etc.)
  * Patient advocates and representatives
  * Researchers in healthcare or technology fields
  * Healthcare administrators and managers
* AIM 1: Must be over 18 years old
* AIM 1: English-speaking
* AIM 1: Willing and able to provide informed consent
* AIM 2 (RURAL OLDER CANCER SURVIVORS): A rural resident based on the Health Resources & Services Administration (HRSA) rural analyzer
* AIM 2 (RURAL OLDER CANCER SURVIVORS): Self-report of diagnosis with any cancer
* AIM 2 (RURAL OLDER CANCER SURVIVORS): Self-report posttreatment (i.e., completion of curative intent therapy including surgery, chemotherapy, molecularly targeted, and endocrine therapy)
* AIM 2 (RURAL OLDER CANCER SURVIVORS): Have access to a computer, a smartphone, or a tablet computer
* AIM 2 (RURAL OLDER CANCER SURVIVORS): Aged > 65 years old
* AIM 2 (RURAL OLDER CANCER SURVIVORS): Assessed as having Cancer and Treatment Distress scale (CTXD) scores > 0.85 at screening
* AIM 2 (RURAL OLDER CANCER SURVIVORS): Have a caregiver willing to participate
* AIM 2 (RURAL OLDER CANCER SURVIVORS): Non-institutionalized
* AIM 2 (RURAL OLDER CANCER SURVIVORS): English proficient
* AIM 2 (RURAL OLDER CANCER SURVIVORS): Willing and able to provide informed consent
* AIM 2 (CAREGIVER): An identified informal caregiver of an eligible ROCS (caregivers include, but are not limited to, a child, partner, or friend; caregivers can reside in a rural or urban area and may or may not live with the ROCS
* AIM 2 (CAREGIVER): Have internet access
* AIM 2 (CAREGIVER): ≥ 18 years old
* AIM 2 (CAREGIVER): Non-institutionalized
* AIM 2 (CAREGIVER): English proficient
* AIM 2 (CAREGIVER): Willing and able to provide informed consent
* AIM 3 (FINAL WORKSHOP): Includes providers, medical and practice managers, patient care coordinators, and medical health technologists

Exclusion Criteria:

* AIM 2 (RURAL OLDER CANCER SURVIVORS): Experience a cancer recurrence or a new cancer diagnosis during their participation in the trial because of the body of literature that reports increased distress associated with cancer recurrence
* AIM 2 (RURAL OLDER CANCER SURVIVORS AND CAREGIVER): Are inpatients
* AIM 2 (RURAL OLDER CANCER SURVIVORS AND CAREGIVER): Cognitive impairment precludes the ability to provide written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 578 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2031-08-26 (Estimated); Study Completion 2032-08-26 (Estimated)

PRIMARY OUTCOMES:
Cancer Related Distress (validated 23-item scale) | Up to 1 year
  Cancer-related distress will be measured using the Cancer and Treatment Distress Scale (23 items; item scores 0-3; higher scores indicate greater distress). The CTXD assesses distress over the past week and includes six subscales: (1) uncertainty, (2) family strain, (3) health burden, (4) finances, (5) identity/appearance, and (6) medical demands. The primary outcome is the mean cumulative score across all items and subscales. A mean score above 0.85 indicates elevated distress in long-term survivors. The CTXD has demonstrated high validity and reliability across time, from pre-treatment to 18 years post-treatment, with Cronbach's alphas ranging from 0.77 to 0.90. The subscales align with the psychosocial domain identified in the NCCN Guidelines for Distress Management.

SECONDARY OUTCOMES:
Self-reported Healthcare Resource Usage | Up to 12 months
  Self-reported healthcare service usage will be measured as a count outcome at 4, 8, and 12 months post-randomization. At each follow-up, participants will report the number of times they accessed healthcare services, including primary care, oncology consultations, mental health counseling, urgent care, and survivorship care visits, since their last assessment. Data will be collected using a structured checklist within the participant survey. Evaluable participants are those who complete the survey. Both service-specific and total counts will be summarized, and a cumulative total across all intervals (0-12 months) will serve as the overall indicator of healthcare resource utilization.
Self-reported Shared Device Use | Up to 12 months
  Assessed as a binary outcome at each follow-up time point (4, 8, and 12 months post-randomization). Participants will report whether they shared a digital device (e.g., smartphone, tablet, or computer) with a caregiver, family member, or friend to access health-related information or services since their last assessment. The structured survey item captures both access and behavioral engagement with health technologies through shared devices.
Telehealth Utilization (self-reported use of portal, completed visits, and visit modality) | Up to 12 months
  Telehealth utilization will be self-reported by rural cancer survivors (ROCS) and caregivers at baseline and follow-up assessments at 4, 8, and 12 months post-randomization. Participants will indicate whether they have used any telehealth services in the last 4 months, and if so, specify the type (e.g., oncology follow-up, primary care, mental health), frequency, and modality (e.g., video, phone).
  Utilization will be operationalized as a binary indicator at each time point (1 = used, 0 = did not use, NA = missing). We will also summarize cumulative utilization across all time points to derive an overall indicator of self-reported telehealth utilization during the 12-month study period.
Cancer Survivors' Unmet Needs (validated 35-item scale) | Up to 12 months
  Cancer Survivors' Unmet Needs will be assessed using a validated 35-item questionnaire evaluating emotional, informational, physical, and practical support needs. A total unmet needs score and domain-specific scores will be calculated per the scoring manual, with higher scores indicating greater levels of unmet need. The outcome will be analyzed as a continuous variable at 4, 8, and 12 months post-randomization. Primary analyses will compare total unmet needs between the CONNECT and control groups at 12 months, with longitudinal models assessing changes across all time points.
Caregiver Strain Index (validated 13-item scale) | Up to 12 months
  Caregiver strain will be measured using the Caregiver Strain Index (CSI), a validated 13-item scale assessing the level of strain experienced by caregivers after hospital discharge of an elderly family member. Each item is scored as 0 (no) or 1 (yes), with total scores ranging from 0 to 13, where higher scores indicate greater caregiver strain. The CSI will be administered at baseline and follow-up assessments (4, 8, and 12 months post-randomization). The outcome will be analyzed as a continuous variable, with the primary comparison of mean CSI scores between the CONNECT and control arms at 12 months to evaluate the cumulative effect of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Marquita W Lewis, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States